CLINICAL TRIAL: NCT00925314
Title: A Phase 2, Open-Label Evaluation of the Safety and Efficacy of CB-10-01, Transgenic Lymphocyte Immunization (TLI) Against Telomerase, as Adjuvant Therapy in Subjects With Stage III Melanoma
Brief Title: A Study of Transgenic Lymphocyte Immunization (TLI) Against Telomerase in Subjects With Stage III Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cosmo Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-10-01-02
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma
Keywords: Stage III Melanoma; Melanoma; TLI; Transgenic Lymphocyte Immunization; CB-10-01-02
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transgenic Lymphocyte Immunization (Experimental): Open Label, Single Arm
  Interventions: Biological: CB-10-01 (Transgenic Lymphocyte Immunization)

INTERVENTIONS:
Biological: CB-10-01 (Transgenic Lymphocyte Immunization) — 1 Primary Infusion and 2 Booster Infusions
  Other Names: TLI

SUMMARY:
The purpose of this study is to assess the safety, efficacy, and immunological response to the study product, TLI, as an adjuvant therapy in subjects with Stage III Melanoma.

Normal cells in the body have an established lifespan. Cancer cells on the other hand have the ability to continue to divide into new cells indefinitely. More than 85% of cancer has this ability because of an enzyme found in the cancer cell. The Investigational Product, Transgenic Lymphocyte Immunization (TLI), is aimed at helping the immune system target this enzyme found in most cancerous cells.

Subjects who meet all inclusion and exclusion criteria will undergo a leukapheresis in which white blood cells will be collected and used to manufacture their own personal study product. Subjects will receive 3 infusions of TLI roughly 1 month apart and will be followed over a 2 year period with routine laboratory draws, computed tomography (CT) scans and physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age and able to understand and give written informed consent
* Women subjects of childbearing potential (WOCBP) and male subjects must be using an effective method of contraception
* Histologic diagnosis of malignant melanoma:

  * Melanoma primary completely resected with negative margins. Primary surgery must be <8 weeks from leukapheresis procedure
  * Stage IIIB or Stage IIIC according to the American Joint Committee on Cancer (AJCC) Tumor-Node-Metastasis (TNM) criteria (Appendix 2) OR previously resected Stage I or II melanoma that recurs as Stage IIIB or IIIC.
* HLA-A2 positive
* ECOG Performance Status of 0, 1 or 2 (Appendix 3)
* Adequate bone marrow, hepatic, and renal function:

  * WBC ≥1500/μL
  * ANC ≥1000/μL
  * Platelets ≥100 × 103/μL
  * Hemoglobin ≥9 g/dL
  * Creatinine ≤2 ULN
  * AST ≤2 ULN
  * Bilirubin ≤2 ULN (except for subjects with Gilbert's Syndrome who must have a total bilirubin <3.0 mg/mL)
* Negative screening tests for HIV, Hepatitis B and C

Exclusion Criteria:

* Female subjects, their partners and male subjects who are unwilling or unable to practice abstinence or use a barrier method (condoms) during intercourse to minimize the risk of exposure to the blood-borne transgene for the entire period of the study and for up to 8 weeks after the last TLI infusion
* Known allergy to DMSO
* Any malignancy from which the subject has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* Primary ocular or mucosal melanoma
* Autoimmune disease: subjects with a documented history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]) that has or may require systemic therapy
* Concomitant therapy with any anticancer agent; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non cancer-related illnesses). Replacement doses of corticosteroids are allowed in subjects with adrenal insufficiency
* Prior biologic therapy for melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the percentage of subjects who have no recurrence of metastatic melanoma at 24 months from the time of primary surgery. | 24 months

SECONDARY OUTCOMES:
Percentage of subjects who have no recurrence of metastatic melanoma 9 and 16 months following the time of primary surgery. | 9 and 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Daniels, MD, PhD, Principal Investigator — University of California, San Diego
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Northern California Melanoma Center, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California